CLINICAL TRIAL: NCT06894537
Title: Efficacy of Echo-guided Percutaneous Electrical Nerve Stimulation of the Femoral Nerve on Explosive Strength and Metabolic Response in Healthy Subjects. A Randomised Clinical Trial.
Brief Title: Echo-guided Percutaneous Electrical Nerve Stimulation of the Femoral Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, PhD, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECO-est
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Health Subjects
Keywords: Percutaneous electrical nerve stimulation; Femoral nerve; Vertical jump; Skin temperature; Physiotherapy
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The intervention of the experimental group will consist of an intervention by performing percutaneous echo-guided electrical nerve stimulation of the femoral nerve.
  Interventions: Other: Experimental (percutaneous echo-guided electrical nerve stimulation)
- Control (Active Comparator): The intervention of the control group will be carried out in the same way as in the experimental intervention, but without increasing the intensity of the current.
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Other: Experimental (percutaneous echo-guided electrical nerve stimulation) — The protocol applied in this study will consist of: 10 stimulations of 10 seconds at 10Hz with a rest of 10 seconds between one stimulation and the next one. The intensity of the current (mA) will be adapted to each of the subjects until the greatest possible muscle contraction is achieved without reaching the painful threshold.
  Arms: Experimental group
Other: Control (placebo) group — For the subjects in the control group, the same process shall be carried out without increasing the intensity of the current. It shall be explained to the subjects that the current will reach a non-perceptible stimulus.
  Arms: Control

SUMMARY:
Introduction. Variables such as pain and strength can be modified in the short and medium term by the application of currents. The percutaneous form of percutaneous needle-guided acupuncture can eliminate the impedance of the surrounding tissues that limit the optimal diffusion of the current to the target tissue. It is necessary to objectify the metabolic response of this technique and its effects in terms of strength and metabolic response.

Objective. To evaluate the safety and efficacy, in acute and subacute phases, of percutaneous electrical nerve stimulation in healthy subjects.

Method. Single-blind randomised clinical study. Thirty-two subjects will be recruited and randomised to the experimental and control groups. The intervention in the experimental group will consist of a percutaneous percutaneous electrical nerve stimulation of the femoral nerve, while in the control group the same intervention will be performed without increasing the intensity of the current. The primary variable will be vertical jump height (My Jump® iOS app) and the secondary variable will be skin temperature (Hikmicro M60 model Hangzhou).

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 18 and 24.
* Of both sexes.
* Who practice sport at least twice a week.
* Who sign the informed consent document.

Exclusion Criteria:

* Medical diagnosis of chronic systemic diseases or diseases that may interfere with thermographic imaging (rheumatoid arthritis, fibromyalgia, deep vein thrombosis, etc.).
* Having undergone lower limb surgery in the 24 months prior to the study.
* Intake of drugs that may influence the thermographic response (antipyretics, non-steroidal anti-inflammatory drugs, topical solutions on the area to be studied, etc.).
* People with nickel allergy or belonephobia (needle phobia).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline jump height after warming, treatment and at 1 and 24 hours | Baseline, within the first seven days after warming, treatment and after 1 and 24 hours follow-up visit
  Using the My Jump® application (iOS app), the jump height is evaluated. This tool measures the time in the air (in milliseconds), indirectly assessing the height of the jump (in centimetres). This tool has shown a high reliability in the evaluation of counter movement jump. The unit of measurement is centimetres (cm), where the higher the centimetres, the higher the jump height.

SECONDARY OUTCOMES:
Change from baseline muscle power after warming, treatment and at 1 and 24 hours | Baseline, within the first seven days after warming, treatment and after 1 and 24 hours follow-up visit
  The metabolic response will be measured with a thermography device (Hikmicro M60 model Hangzhou camera). This complementary imaging technique analyses infrared radiation emitted by object surfaces (skin) and reflects the state of molecular agitation, providing objective information on the metabolic state of the underlying structures. The assessment shall be performed according to the consensus document on control variables in thermographic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No